CLINICAL TRIAL: NCT01622556
Title: Phase II Trial of Reduced Intensity Conditioning (RIC) and Allogeneic Transplantation of Umbilical Cord Blood (UCB) From Unrelated Donors in Patients With Hematologic Malignancies
Brief Title: Conditioning Treatment With Umbilical Cord Blood Transplant for Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Amer Beitinjaneh, MD, Assistant Professor of Medicine, Medical Director Stem Cell Transplant Unit, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15954 UCB-2011
Record Dates: First submitted 2012-06-08; First posted 2012-06-19 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Hematologic Malignancies
Keywords: Chronic Myeloid Leukemia; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Non-Hodgkins Lymphoma; Hodgkin's Disease; Myelodysplastic Syndromes; Myeloproliferative Disorder
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — fludarabine; Busulfan; thymoglobulin; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced Intensity Conditioning with UCB Transplant (Experimental)
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Thymoglobulin; Radiation: Total Body Irradiation; Biological: Umbilical Cord Blood

INTERVENTIONS:
Drug: Fludarabine — 35 mg/m2 IV/day x 5 days
Drug: Busulfan — .8 mg/kg IV Q6h x 8 doses
Drug: Thymoglobulin — 1.5 mg/kg/day x 3 days
Radiation: Total Body Irradiation — 150 cGy for 2 days
Biological: Umbilical Cord Blood — Two partially HLA-matched UCB units. Each unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient.

SUMMARY:
This is a phase II study to assess the day 180 event free and overall survival after administration of a specified combination of fludarabine, busulfan, Total Body Irradiation (TBI), and thymoglobulin reduced intensity conditioning and 2 unit UCB stem cell transplant in a single institution setting in patients with hematologic malignancies for whom allogeneic transplantation is indicated.

ELIGIBILITY:
Inclusion Criteria:

Subjects 18-70 years old. ECOG 0-2

Patients must have a diagnosis of one of the following:

* Chronic Myeloid Leukemia
* Acute Myeloid Leukemia
* Acute Lymphoblastic Leukemia
* Hodgkin's Disease
* Non-Hodgkins Lymphoma
* Myelodysplastic Syndromes
* Myeloproliferative Disorder

Patients must have adequate visceral organ function

* Patients must furnish written informed consent and HIPAA authorization for release of personal health information.
* Patients must be able to understand the requirements of the study, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

* Patients who have a histocompatible sibling-matched donor age 18 to 65 years in good health who is willing to donate stem cells are ineligible.
* Patients who are pregnant are ineligible.
* Patients are ineligible if they have received cumulative chemotherapy doses in excess of: carmustine (BCNU) 400 mg/m2, and/or a cumulative anthracycline exposure in excess of 550 mg/m2 doxorubicin (Adriamycin®) unless gated-pool radionuclide cardiac scan shows greater than/equal to 45% ejection fraction.

Patients who are HIV or HTLV-I, -II antibody sero-positive are ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 180 days
  Number of subjects surviving with no events at 180 days post transplantation (Day 0).

SECONDARY OUTCOMES:
Transplant Engraftment | Day 42
  Number of patients with successful UCB engraftment.
Incidence of Graft-versus-host disease (GVHD) | 1 year
  Number of patients that experience acute or chronic GVHD.
Time course for peripheral blood chimerism. | 56 days
  Percent of patients with >95% donor chimerism.
Incidence of secondary lymphoproliferative diseases | 6 months
  Number of patients with secondary lymphoproliferative diseases.
Incidence of disease recurrence | Up to two years
  Number of patients experience disease recurrence.
Incidence of serious infectious complications | 1 year
  Number of patients experiencing serious infectious complications.
Overall Survivals | 60 months
  Number of patient with overall event free survival and overall survival distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Beitinjaneh, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States